CLINICAL TRIAL: NCT02362828
Title: EPiMAP Obstetrics: European Practices in the Management of Accidental Dural Puncture in Obstetrics: European Prospective Multicentre Observational Audit to MAP Out Current Practices in the Management of Patients Who Had Accidental Dural Puncture During EPIdural Insertion
Brief Title: EPiMAP Obstetrics: European Practices in the Management of Accidental Dural Puncture in Obstetrics
Acronym: EPiMAP
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: EPiMAP Obstetrics
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2018-12

CONDITIONS: Post-Dural Puncture Headache
Keywords: Post-Dural Puncture Headache; Blood Patch, epidural; Obstetrics; European Society of Anaesthesiology (ESA); epidemiology; Accidental Dural Puncture (ADP); Anaesthesia; childbirth complication; epidural analgesia; postdural puncture headache; prophylactic epidural blood patch; epidural
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of EPiMAP Obstetrics are:

* to identify risk factors for failure of epidural blood patch in the obstetric population for management of post dural puncture headache.
* to describe European practices in the management of accidental dural puncture in the Obstetric population.

DETAILED DESCRIPTION:
The primary aim of this prospective, international audit of practice is to identify risk factors for failure of epidural blood patch (EBP) in the Obstetric population after accidental dural puncture (ADP) with an epidural needle. Other aims are to describe the epidemiology, management principles, side effects and complications of ADP and longer-term effects of ADP on patients undergoing Obstetric anaesthesia and analgesia. Expectation is that this audit of practice will provide important information in understanding the reasons for failure of EBP and subsequently to better manage parturients affected by this debilitating complication.

Postdural puncture headache (PDPH) is the most common serious complication of accidental dural puncture (ADP), and feared by every Anaesthesiologist. It is associated with significant peri-partum maternal distress, and poor bonding with the baby, which in turn leads to physical disability for the mother and psychological and social implications for the whole family. It is estimated that about 10,000 parturients in Europe may have an accidental dural puncture (ADP) each year. Attitudes and practices in the management of ADP are based on small studies, and sometimes driven by experience rather than evidence. Although several methods have been described in the literature to treat PDPH, one common method used is an epidural blood patch (EBP). This is believed to be successful in about 60-80% of parturients on the first attempt, but results from most studies are based on a small numbers of patients. The reasons and predisposing factors for success and failure of different management strategies, specifically EBP, therefore needs to be investigated and described. Large observational studies on post-dural puncture headache in the Obstetric population are singularly absent from the literature.

ELIGIBILITY:
Inclusion Criteria:

* All women ≥ 18 years old, who develop classical symptoms of post-dural puncture headache after epidural anaesthesia for labour or for caesarean section.

Exclusion Criteria:

* Post-dural puncture headache following deliberate dural puncture with a spinal needle in women where there was no observed accidental dural puncture with an epidural needle.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women ≥ 18 years old, who develop classical symptoms of post-dural puncture headache after epidural anaesthesia for labour or for caesarean section.
Sampling Method: Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
To examine the risk factors for failed epidural blood patch (EBP) following post-dural puncture headache | 24 h after application of Epidural blood patch
  To examine the risk factors for failed epidural blood patch (EBP) following post-dural puncture headache, in the obstetric population. Failure would be defined as lack of reduction in pain intensity by at least 50% at 24 h after application of EBP, compared to worst pain before EBP or a visual analogue pain score (VAS pain) of > 3 at 24 h.

SECONDARY OUTCOMES:
European practices in the management of Post Dural Puncture Headache (PDPH) | 24 h after application of Epidural blood patch
Incidence of significant Post Dural Puncture Headache (PDPH) and treatment failure in different countries in Europe | 24 h after application of Epidural blood patch
Timing of the procedure (after diagnosis of PDPH) and the volume of blood injected in relation to success or failure | 24 h after application of Epidural blood patch
Complications and side effects of Epidural blood patch (EBP) | 24 h after application of Epidural blood patch
  Complications include : Chronic headache and backache, neurological injuries, audiological or visual other chronic impairments
Variation in practices for management of Accidental Dural Puncture (ADP) in different European countries | 24 h after application of Epidural blood patch

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gupta, MD, Study Chair — Karolinska University Hospital
Locations (1):
- Karolinska Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Gupta A, von Heymann C, Magnuson A, Alahuhta S, Fernando R, Van de Velde M, Mercier FJ, Schyns-van den Berg AMJV; EPiMAP collaborators. Management practices for postdural puncture headache in obstetrics: a prospective, international, cohort study. Br J Anaesth. 2020 Dec;125(6):1045-1055. doi: 10.1016/j.bja.2020.07.061. Epub 2020 Oct 8. PMID 33039123
- [Derived] Gupta A, Van de Velde M, Magnuson A, von Heymann C, Guasch E, Alahuhta S, Mercier FJ, Schyns-van den Berg AMJV; European Practices in the Management of Accidental Dural Puncture in Obstetrics Investigators. Factors associated with failed epidural blood patch after accidental dural puncture in obstetrics: a prospective, multicentre, international cohort study. Br J Anaesth. 2022 Nov;129(5):758-766. doi: 10.1016/j.bja.2022.06.040. Epub 2022 Sep 3. PMID 36064491